CLINICAL TRIAL: NCT02936063
Title: Outcomes Comparing Different Methods of Skin Closure in Patients Undergoing Head and Neck Surgery.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left the institution before any participants were enrolled.
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-34701
Record Dates: First submitted 2016-06-29; First posted 2016-10-18 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Surgical Wound
Keywords: Head and neck surgery; Scar cosmesis; Surgical staples; Sutures; Patient satisfaction
MeSH Terms: conditions — Surgical Wound; Patient Satisfaction | interventions — Sutures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical staples (Experimental): Skin closure with surgical staples
  Interventions: Procedure: Surgical staples
- Sutures (Experimental): Skin closure with subcuticular sutures
  Interventions: Procedure: Subcuticular sutures

INTERVENTIONS:
Procedure: Surgical staples — Closure of surgical wound at skin level with surgical staples
  Arms: Surgical staples
Procedure: Subcuticular sutures — Closure of surgical wound at skin level with subcuticular sutures
  Arms: Sutures

SUMMARY:
When patients undergo neck dissection surgeries, the current standard of care is to close the skin layer with either metal staples, which are removed a few days post-operatively, or with sutures, which can be absorbable or removed. To date, there is no conclusive data in the literature that definitively suggests one method is better than the other, with regard to wound complications or mature scar cosmesis. Currently, skin closure method is chosen by each individual surgeon, and is based on personal preference, factoring in evaluation of the wound. The goal of the study is to compare the two methods of skin closure, and the measured outcomes the investigators will be looking at are patient satisfaction, wound complications, and mature scar cosmesis. The investigators will be randomizing patients undergoing head and neck surgery to receive either staples or subcuticular sutures, and giving them surveys at their post-operative clinic visits to evaluate the outcomes, to determine if patients perceive one method to be superior to the other.

DETAILED DESCRIPTION:
The goal of the study is to evaluate and compare patient perception of two different methods of skin closure following head and neck surgery. Currently, the standard of care includes closing with surgical staples or subcuticular sutures, and is decided at surgeon's discretion. Both methods are used in accordance with the standard of care at Boston Medical Center, depending on individual physician preference. There are also factors that may influence choice of closure at time of surgery, such as operative time, or wound characteristics. For instance, if the operative time was already extending longer than expected, to decrease patient anesthesia time, the surgeon may opt for staples, since they are faster to place than sutures. Also, although a rare scenario, if there was excessive blood loss during the surgery or the surgeon has reason to suspect post-operative hematoma development, they will likely opt for staple closure, to facilitate easy post-operative access to the wound if necessary. In the literature, incidence of hematoma as a post-operative complication to head and neck surgery is stated as 3-4.7%.

There have been various studies in the literature comparing these two skin closure methods for general surgery (abdominal procedures) and obstetrics/gynecological surgeries, with inconclusive outcomes. We found a lack of data in the literature describing head and neck surgeries. Given the different type of wounds, and the often more visible nature of the resulting scars, the investigators believe there is value to accessing patient perception of skin closure in this cohort. Kobayashi et al. conducted a large randomized control trial of 1264 subjects, comparing staples vs. subcuticular sutures after open and laparoscopic elective colorectal cancer surgery. The results of the study showed no significant difference in operative outcomes (wound complications, surgical site infections, post-operative length of stay, scar esthetics). However, staples were found to have a shorter operative time, while sutures resulted in statistically significant higher patient satisfaction. A meta-analysis of 12 studies comparing sutures and staples in caesarian section showed no difference in patient satisfaction or scar cosmesis, but found more wound complications in the staples arm. Much of the existing data are reported from general surgery or obstetrics/gynecology. There is not a lot of literature in otolaryngology or head and neck surgery that evaluates skin closure methods. The importance of cosmetic outcomes and patient satisfaction is particularly important in the field of head and neck surgery, due to the visibility of the scars given their location.

Upon review of the existing literature, there is no definitive data to support either method as superior, with regards to wound complications and outcomes, mature scar cosmesis, or post-operative pain. There is some evidence to suggest that subcuticular suture closure is marginally superior with regards to scar cosmesis, but given that operative time is increased, there is not enough benefit to the patient to change the standard of care. In addition, with the current trend of medicine moving towards patient-reported outcomes, it becomes increasingly important to evaluate patient satisfaction to determine whether there is a superior method. The investigators hypothesize that there will be no statistically significant difference between staple skin closure and subcuticular suture closure, with regards to the primary outcomes of patient satisfaction and mature scar cosmesis.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide informed consent
* Ability to speak/read English language
* Adult patients (age > 18)
* Willing to have follow-up appointments (per clinical care protocol)
* Both genders

Exclusion Criteria:

* Prior radiation therapy to the head and neck region (prior to surgery)
* Prior surgery to the head and neck region (at the judgement of investigator)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03 (Estimated); Primary Completion 2019-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Patient and Observer Scar Assessment Survey (POSAS) | 2 years post-operative
  Survey score - to assess for scar cosmesis outcome

SECONDARY OUTCOMES:
Patient Satisfaction Survey | 2 years post-operative
  Survey score - to assess for patient satisfaction
Wound complications - dehiscence | 2 years post-operative
  Wound dehiscence
Wound complications - infection | 2 years post-operative
  Surgical site infections

CONTACTS AND LOCATIONS:
Overall Officials: Scharukh Jalisi, MD, MA, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No